CLINICAL TRIAL: NCT00024115
Title: Phase I Study of Recombinant BL22 Immunotoxin in Patients With CD22-Positive B-Cell Non-Hodgkin's Lymphoma or Chronic Lymphocytic Leukemia
Brief Title: BL22 Immunotoxin in Treating Patients With Non-Hodgkin's Lymphoma or Chronic Lymphocytic Leukemia
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068892; NCI-01-C-0213; NCI-5336; NCT00021593 (obsolete NCT alias)
Record Dates: First submitted 2001-09-13; First posted 2003-01-27 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2006-12

CONDITIONS: Leukemia; Lymphoma
Keywords: refractory chronic lymphocytic leukemia; B-cell chronic lymphocytic leukemia; stage III grade I follicular small cleaved cell lymphoma; stage III grade II follicular mixed cell lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage IV grade I follicular small cleaved cell lymphoma; stage IV grade II follicular mixed cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; recurrent grade I follicular small cleaved cell lymphoma; recurrent grade II follicular mixed cell lymphoma; recurrent grade III follicular large cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult diffuse small noncleaved cell/Burkitt's lymphoma; prolymphocytic leukemia; contiguous stage II grade I follicular small cleaved cell lymphoma; contiguous stage II grade II follicular mixed cell lymphoma; contiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II grade I follicular small cleaved cell lymphoma; noncontiguous stage II grade II follicular mixed cell lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; stage III diffuse small lymphocytic/marginal zone lymphoma; contiguous stage II diffuse small lymphocytic/marginal zone lymphoma; noncontiguous stage II diffuse small lymphocytic/marginal zone lymphoma; stage IV diffuse small lymphocytic/marginal zone lymphoma; recurrent diffuse small lymphocytic/marginal zone lymphoma; recurrent mantle cell lymphoma
MeSH Terms: conditions — Leukemia; Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Prolymphocytic; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Mantle-Cell | interventions — RFB4(dsFv)-PE38 recombinant immunotoxin; Immunization, Passive; Adjuvants, Immunologic

INTERVENTIONS:
Drug: BL22 immunotoxin
Procedure: antibody therapy
Procedure: biological response modifier therapy
Procedure: immunotoxin therapy

SUMMARY:
RATIONALE: The BL22 immunotoxin can locate tumor cells and kill them without harming normal cells.

PURPOSE: Phase I trial to study the effectiveness of the BL22 immunotoxin in treating patients who have non-Hodgkin's lymphoma or chronic lymphocytic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the toxicity and therapeutic efficacy of recombinant BL22 immunotoxin in patients with CD22-positive B-cell non-Hodgkin's lymphoma or chronic lymphocytic leukemia.
* Determine the pharmacokinetics, including the terminal elimination serum half-life area under the curve and volume of distribution, of recombinant BL22 immunotoxin in these patients.
* Determine the immunogenicity of recombinant BL22 immunotoxin in these patients.
* Determine the effect of recombinant BL22 immunotoxin on various components of the circulating cellular immune system in these patients.

OUTLINE: This is a dose-escalation study.

Patients receive recombinant BL22 immunotoxin IV over 30 minutes on days 1, 3, and 5. Patients may be retreated at least every 20 days for up to 25 courses in the absence of disease progression and sufficient neutralizing antibodies.

Cohorts of 3-6 patients receive escalating doses of recombinant BL22 immunotoxin until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity.

PROJECTED ACCRUAL: A total of 40 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed chronic lymphocytic leukemia or prolymphocytic leukemia:
* Failed prior standard chemotherapy and treatment is medically indicated as evidenced by the following:
* Progressive disease-related symptoms
* Progressive cytopenias due to marrow involvement
* Progressive or painful splenomegaly or adenopathy
* Rapidly increasing lymphocytosis
* Autoimmune hemolytic anemia or thrombocytopenia
* Increased frequency of infections OR
* Confirmed CD22+ B-cell indolent non-Hodgkin's lymphoma
* Stages II-IV that have failed at least 1 prior standard therapy and treatment is medically indicated
* No patients whose serum neutralizes BL22 or PE38 in tissue culture, due to antitoxin or antimouse-IgG antibodies
* No central nervous system disease requiring treatment
* If the patient is non-leukemic, the absolute neutrophil count must be greater than 1,000/mm3 and the platelet count greater than 40,000/mm3

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 60-100%

Life expectancy:

* More than 6 months

Hematopoietic:

* See Disease Characteristics

Hepatic:

* ALT and AST less than 5 times upper limit of normal

Renal:

* Adequate renal function

Pulmonary:

* Adequate pulmonary function

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* HIV negative

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Prior bone marrow transplantation allowed
* At least 3 weeks since prior interferon for malignancy

Chemotherapy:

* See Disease Characteristics
* At least 3 weeks since prior cytotoxic chemotherapy for malignancy

Endocrine therapy:

* Not specified

Radiotherapy:

* At least 3 weeks since prior radiotherapy for malignancy

Surgery:

* Not specified

Other:

* At least 3 weeks since prior retinoids
* At least 3 weeks since prior systemic therapy for cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Kreitman, MD, Study Chair — National Cancer Institute (NCI)
Locations (1):
- Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland, United States